CLINICAL TRIAL: NCT06247371
Title: Randomised Controlled Trial of a Heart Failure Medication Decision Aid in Singapore
Brief Title: Impact of a Novel Heart Failure Medication Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ng Teng Fong General Hospital (Other)
Responsible Party: Principal Investigator, Shen Qianyu, Researcher, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/00772
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Randomised controlled trial; Decision aid; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: This study incorporates a prospective single centre, two arms parallel randomised controlled trial with 1:1 patient allocation.
Who Masked: Participant
Masking Description: Only participants are masked to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid (Experimental): Patients will be presented with a decision aid featuring personalized cost information, as well as other information about angiotensin receptor neprilysin inhibitor (ARNI) and angiotensin-converting enzyme inhibitor (ACEI) medications. These patients will then be tasked to choose a preferred medication and reflect on which attribute holds the most significance for them. The preferred medication will be communicated to the clinicians during the clinic session.
  Interventions: Behavioral: Decision aid
- Usual care (No Intervention): Patients are managed as per usual clinical routine without the decision aid.

INTERVENTIONS:
Behavioral: Decision aid — The Singapore developed HF DA is a A3 sized one-page poster designed to convey information about HF medications options (ACEI and ARNI only) and their pros and cons. The DA contains informative attributes of both medications that are presented side by side for comparison. These attributes include subsidized cost, frequency of use, duration of use, route of administration, low blood pressure side effect rate and benefits such as non-hospitalization rate and survival rate.
  Arms: Decision aid

SUMMARY:
A modified Zelen design randomised controlled trial over 6 months period is designed to investigate the influence of a heart failure medication decision aid prior to clinic session on shared decision making and its long term effect. Participants are randomised to either the decision aid arm or the usual care arm.

DETAILED DESCRIPTION:
A novel heart failure (HF) medication decision aid (DA) has been constructed, taking into account the needs of both patients and clinicians. Developed with a focus on brevity, this single-page DA is designed to offer patients a quick and concise overview of the information they desire about their medication ahead of their clinic session. It encompasses personalised cost information, considering the subsidies available in Singapore. The aim of the DA is to improve the communication between clinicians and HF patients. The conduct of this randomized controlled trial (RCT) is to study the effectiveness of the HF DA in the real-world setting.

Patients are randomized to either the DA arm or the usual care (UC) arm. In the DA group, patients will be provided with a DA featuring duration and frequency of use, benefits, side effect and cost information about angiotensin receptor neprilysin inhibitor and angiotensin-converting enzyme inhibitor medications. These patients will then be tasked to choose a preferred medication and reflect on which attribute holds the most significance for them. The preferred medication will be communicated to the clinicians during the clinic session. For the UC arm, clinicians will manage the encounter as per current usual routine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure with reduced ejection fraction (HFrEF)
* Singaporean nationality

Exclusion Criteria:

* Patient is currently on Medifund OR have Medical Claims Pro-ration System (MCPS)
* Pregnant
* Age 21 years and below
* Incapable of personally giving consent
* Unable to speak and read English or Chinese

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Frequency of Medication cost discussion | Day 1 (Clinic session)
  This outcome will be measured using an audio recording of the clinic session. Audio recording will be transcribed. The presence of cost discussion during the clinic session will coded based on Hunter et al. (2016) definition. Presence of cost discussion is coded as 1 and absence of cost discussion is coded as 0. Coding of cost discussion frequency will be done by 2 analysts who are blinded to the randomisation.

SECONDARY OUTCOMES:
Decisional conflict | Day 1 (Immediately after clinic session) and Day 180 (Follow-up appointment)
  Decisional conflict is defined as uncertainty when faced with choosing among competing options that can impact patient's personal values or well-being. The Decisional Conflict Scale (DCS) contains 16 items with 5 responses. The level of decisional conflict is reported from 0 to 100, with 0 indicating a high degree of certainty about the best choice and 100 indicating a significant degree of uncertainty about the best choice.
Decision satisfaction | Day 1 (Immediately after clinic session) and Day 180 (Follow-up appointment)
  Patient's satisfaction with their decision will be measured with the Satisfaction with Decision Scale (SWD) developed by Holmes-Rovner. The SWD is a reliable tool consisting of 6 items. Respondents rate each item on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree." A higher score indicates greater decisional satisfaction.
Decision regret | Day 180 (Follow-up appointment)
  The Decision Regret Scale (DRS) evaluates the degree of regret that an individual experiences after making a decision. DRS has demonstrated strong internal consistency and includes five items. A score of 0 suggests the absence of any regret, while a score of 100 indicates a high level of regret.
Prescribed medication agreement with preferred medication | Day 1 (Immediately after clinic session)
  Patient's prescribed medication record will be obtained from the electronic medical record. Their preferred medication choice will be documented after reading the decision aid. Presence of agreement is coded as 1 and presence of discrepancy is coded as 0.
Health-related quality of life | Day 1 (Immediately after clinic session) and Day 180 (Follow-up appointment)
  Patients will assess their HRQoL with EuroQol scale (EQ-5D-5L). The EQ-5D-5L score is calculated using a standardized algorithm that considers five dimensions (mobility, self-care, usual activities, pain, and anxiety/depression). Each dimension has five response levels (no problems, slight problems, moderate problems, severe problems or extreme problems). The algorithm produces a level sum score that ranges from 5 to 25 with 25 being the worst health and 5 being perfect health.
Financial toxicity | Day 1 (Immediately after clinic session) and Day 180 (Follow-up appointment)
  Patient's financial well-being will be assessed with COST-FACIT questionnaire. The questionnaire contains twelve items with a total score of 0 to 44. The higher the score, the better the financial well-being. The threshold for financial toxicity is defined as a score < 26.
Readmission rate | Day 180 (Follow-up appointment)
  Electronic medical record will be used to evaluate this outcome measures. The frequency of readmission into hospital within 6 months of recruitment will be tallied and compared between arms.
Heart Failure symptoms and Adverse drug reactions | Day 180 (Follow-up appointment)
  Clinician's notes will be used to evaluate these two outcome measures. The frequency of various heart failure symptoms and drug reactions will be tallied within 6 months of recruitment and compared between arms.
Medication Adherence | Day 180 (Follow-up appointment)
  Medication adherence will be captured by generating the Medication Possession Ratio using the pharmacy database. The higher the ratio, the better the medication adherence. The ratio between the two arms will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Hwee Lin Wee, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Ng Teng Fong General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for sharing upon request.
Supporting Information: Study Protocol
Time Frame: Supporting information and IPD will be made available after publication of trial results
Access Criteria: Data will be made available for sharing upon request, after execution of a data sharing agreement.